CLINICAL TRIAL: NCT02846896
Title: The Health Burden of Primary Biliary Cirrhosis (PBC) in Switzerland
Status: Completed | Type: Observational
Sponsor: Fondazione Epatocentro Ticino (Other)
Collaborators: Vifor Pharma (Industry); Intercept Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: SwissPBC - SASL36
Record Dates: First submitted 2016-07-25; First posted 2016-07-27 (Estimated); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Primary Biliary Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis, Biliary

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
PBC is a rare, autoimmune, cholestatic liver disease with genetic and environmental pathogenetic factors. Data about epidemiology of PBC in Switzerland are completely lacking. Epidemiology can be a powerful tool in yielding important clues as to burden and etiology of diseases. In addition, the investigators study will be the first one carried out in the country on PBC, and therefore will raise disease awareness and create a network.

ELIGIBILITY:
Inclusion Criteria:

* PBC patients living in Switzerland

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PBC patients living in Switzerland
Sampling Method: Non-Probability Sample
Enrollment: 501 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Prevalence of PBC in Switzerland | from 1.1.2005 until 31.12.2015

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Epatocentro Ticino, Lugano, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Terziroli Beretta-Piccoli B, Stirnimann G, Cerny A, Semela D, Hessler R, Helbling B, Stickel F, Kalid-de Bakker C, Bihl F, Giostra E, Filipowicz Sinnreich M, Oneta C, Baserga A, Invernizzi P, Carbone M, Mertens J. Geoepidemiology of Primary Biliary Cholangitis: Lessons from Switzerland. Clin Rev Allergy Immunol. 2018 Apr;54(2):295-306. doi: 10.1007/s12016-017-8656-x. PMID 29181702